CLINICAL TRIAL: NCT03009448
Title: The Experience of Older Adults Facing Depression for the First Time in Old Age
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: shalvataMHC
Record Dates: First submitted 2016-12-23; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: MAjor Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Late onset depression
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Each subject will be interviewed using a semi constructed interview.

SUMMARY:
Analysis of recent studies show that researchers find it hard to distinguish between Late Onset Depression, a first diagnosed major depressive episode which occurs at old age, and Early Onset Depression, a depressive episode at old age with a history of previous episodes. Since current data, about the phenomenology and etiology of Late Onset Depression, lake conicity it is unclear whether this phenomena should be considered as a distinct subtype of depression. Nevertheless, the wide spread assumption is that Late Onset Depression has a stronger correlation with brain damage and environmental risk factors such as the common losses at old age and weaker correlation with family history and genetics when compared to Early Onset. Although many researchers consider brain damage to have the main contribution to the emerge of Late Onset Depression, the fact that depression has a negative effect on one's health supports the claim that it might be the result and not the rick factor. Since Late Onset Depression correlates with the common losses at old age, the investigators propose that an existential approach that deals with one's meaning, freedom, responsibly and death, might be more appropriate. Thus, the investigators ask how do older adults experience depression which they face for the first time in old age? Current study will seek to understand older adults' experience of Late Onset depression through existential paradigm by using a semi constructed interview.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 67 or more, women aged 62 or more
2. Diagnosis of Major Depressive Disorder, Minor Depressive Disorder or Adjustment Disorder with depressive features made after the age of 67 with men and 62 with women.
3. Basic understanding and ability to converse in Hebrew.

Exclusion Criteria:

1. History of at least one previous major depressive or minor depressive episode before the age of 62 with women or 67 with men
2. Mental Retardation or Autistic Spectrum Disorder
3. Significant cognitive impairment observed by the primary physician.
4. Schizophrenia or Schizoaffective disorder.
5. Depressive episode with psychotic features
6. Substantial suicidality

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Israeli men and women after the age of retirement, 67 and 62 respectably, who are diagnosed with a major depressive episode, minor depressive episode or show depressive symptoms for the first time in their lives at old age.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Data analysis | 10 weeks
  All the data collected, from each semi structured interview, will be analyzed by the investigator to find similarities or differences between the older adults' experience and to identify specific existential themes.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel